CLINICAL TRIAL: NCT02325999
Title: Endoscopic Submucosal Dissection Combine With Laparoscopic Regional Lymph Node Dissection:a New Therapy for Early Gastric Cancer
Brief Title: Endoscopic Submucosal Dissection Combine With Laparoscopic Regional Lymph Node Dissection for Early Gastric Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hua Meng, Endoscopic Submucosal Dissection combine with Laparoscopic Regional Lymph node Dissection for early gastric cancer, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESDLD2013; BeijingFHMH2013 (Other Grant/Funding Number: BeijingFH)
Record Dates: First submitted 2013-12-31; First posted 2014-12-25 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Early Gastric Cancer
Keywords: Endoscopic Submucosal Dissection; Laparoscopic Regional Lymph node Dissection; early gastric cancer; Disease-free survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — s-formylglutathione hydrolase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESD and LRLD (Experimental): The experimental group accept Endoscopic Submucosal Dissection Combine With Laparoscopic Regional Lymph Node Dissection.
  Interventions: Procedure: ESD AND LRLD
- Endoscopic Submucosal Dissection (ESD) (No Intervention): The group accept Endoscopic Submucosal Dissection only.

INTERVENTIONS:
Procedure: ESD AND LRLD — A new therapy for gastric cancer : Endoscopic Submucosal Dissection combine with Laparoscopic Regional Lymph node Dissection.
  Arms: ESD and LRLD

SUMMARY:
The purpose of this study is to determine whether Endoscopic Submucosal Dissection combine with Laparoscopic Regional Lymph node Dissection for early gastric cancer can improve Disease-free survival ？

DETAILED DESCRIPTION:
Patients with early stage of gastric cancer(T1a/T1bN0M0,NCCN2014.V1) will depart into two group randomized double-blind, then experimental group accept Endoscopic Submucosal Dissection combine with Laparoscopic Regional Lymph node Dissection ,and control group accept Endoscopic Submucosal Dissection only.The follow-up time is from operation to recrudescence.

ELIGIBILITY:
Inclusion Criteria:

* cT1a：ulcer（+）and lesion diameter>3cm and differentiated type. Any ulcer and lesion diameter d>2cm and poorly differentiated type.
* cT1b: Submucosal injection (+)

Exclusion Criteria:

* metastasis
* recrudescence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
DFS | Five years
  Follow-up Disease-free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Shu-tian ZHANG, Study Chair — Beijing Friendship Hospital
Locations (1):
- The capital health research and development of special, Beijing, Beijing Municipality, China